CLINICAL TRIAL: NCT07221032
Title: Phase I Study of FT836 CAR T-cell Therapy in Combination With Daratumumab in Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: FT836 CAR T-cell Therapy in Combination With Daratumumab in Patients With Relapsed and/or Refractory Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Binod Dhakal, Associate Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IIT-DHAKAL-FT836-DARA
Record Dates: First submitted 2025-10-23; First posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Relapse Multiple Myeloma; Refractory Multiple Myeloma
Keywords: multiple myeloma; CAR-T therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- FT836 CAR T cells (1 x 10^8 cells per dose) (Experimental): This is Dose Level 0 (de-escalation dose).
  Interventions: Biological: FT836 CAR T cells (1 x 10^8 cells per dose); Drug: Daratumumab 16 mg/kg
- FT836 CAR T cells (3 x 108 cells per dose) (Experimental): This is Dose Level 1 (starting dose).
  Interventions: Biological: FT836 CAR T cells (3 x 108 cells per dose); Drug: Daratumumab 16 mg/kg
- FT836 CAR T cells (up to 9 x 108 cells per dose) (Experimental): This is Dose Level 2, which is ≤3 times Dose Level 1.
  Interventions: Biological: FT836 CAR T cells (up to 9 x 108 cells per dose); Drug: Daratumumab 16 mg/kg

INTERVENTIONS:
Biological: FT836 CAR T cells (1 x 10^8 cells per dose) — FT836 CAR T cells will be administered by IV injection.
  Arms: FT836 CAR T cells (1 x 10^8 cells per dose)
Biological: FT836 CAR T cells (3 x 108 cells per dose) — FT836 CAR T cells will be administered by IV injection.
  Arms: FT836 CAR T cells (3 x 108 cells per dose)
Biological: FT836 CAR T cells (up to 9 x 108 cells per dose) — FT836 CAR T cells will be administered by IV injection.
  Arms: FT836 CAR T cells (up to 9 x 108 cells per dose)
Drug: Daratumumab 16 mg/kg — Daratumumab will be administered intravenously.
  Other Names: DARZALEX

SUMMARY:
This is a phase I, interventional, single-arm, open-label, dose-finding treatment study designed to evaluate the safety and preliminary efficacy of FT836 in combination with daratumumab in adult patients with relapsed and/or refractory myeloma who have failed prior therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must ≥18 years and < 80 years old.
2. Patients must have received >=3 prior lines of therapies, including proteasome inhibitor, immunomodulator and a CD38 monoclonal antibody:

   • International Myeloma Working Group (IMWG) criteria define refractory disease as disease progression on or within 60 days of receiving therapy.
3. Patients must have measurable disease, including at least one or more of the following criteria:

   1. Serum M-protein ≥ 0.5 g/dl;
   2. Urine M-protein ≥ 200 mg/24 hrs;
   3. Involved serum light chain ≥100 mg/L with abnormal light chain ratio;
4. Karnofsky performance score ≥70.
5. Adequate hepatic function, defined as:

   1. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase <3x upper limit of normal (ULN);
   2. Serum bilirubin <2.0 mg/dL except for patients with Gilbert's syndrome, who must have serum bilirubin of <3 mg/dL.
6. Absolute neutrophil count (ANC) ≥1,000 with no G-CSF within 72 hours or pegylated G-CSF within 10 days.
7. Platelets ≥50,000 with no transfusion within 72 hours of eligibility testing.
8. Adequate renal function, defined as creatinine clearance ≥50 mL/min calculated using the Cockroft-Gault formula.
9. Able to provide written informed consent.
10. Agree to practice birth control during the study.
11. Adequate cardiac function as indicated by New York Heart Association (NYHA) classification I or II AND left ventricular ejection fraction of ≥45% -- by cardiac echocardiogram (ECHO) or multigated acquisition scan (MUGA) -- and adequate pulmonary function as indicated by room air oxygen saturation of ≥90%.
12. Expected survival >12 weeks.
13. Negative urine or serum pregnancy test in females of childbearing potential at study entry.
14. No contraindication to central line access. Female subjects of reproductive potential (women who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months, or have not undergone a sterilization procedure [hysterectomy or bilateral oophorectomy]) must have a negative serum or urine pregnancy test performed as part of the eligibility criteria. Lactating women are eligible for this study but will be asked not to provide breast milk to their child from Day -11 through Day +90 after CAR T-cell therapy. It is possible they may no longer be able to lactate after receiving chemotherapy and treatment.

Due to the high-risk level of this study, while enrolled, all subjects must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization). Additionally, if participating in sexual activity that could lead to pregnancy, the study subject must agree to use reliable and double-barrier methods of contraception during the follow-up period of the protocol.

Acceptable birth control includes a combination of two of the following methods:

* Condoms (male or female) with or without a spermicidal agent.
* Diaphragm or cervical cap with spermicide.
* Intrauterine device (IUD).
* Hormonal-based contraception. Subjects who are not of reproductive potential (women who are premenarche or have been post-menopausal for at least 24 consecutive months or have undergone hysterectomy, tubal ligation, salpingectomy, and/or bilateral oophorectomy or men who have documented azoospermia) are eligible without requiring the use of contraception.

Exclusion Criteria:

1. Positive beta-Human Chorionic Gonadotropin (HCG) in female of child-bearing potential.
2. Confirmed active human immunodeficiency virus (HIV), Hepatitis B or C infection.
3. History of significant autoimmune disease OR active, uncontrolled autoimmune phenomenon requiring steroid therapy defined as >20 mg of prednisone or equivalent daily.
4. Presence of ≥ Grade 3 non-hematologic toxicities as per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 from any previous treatment unless it is felt to be due to underlying disease.
5. Concurrent use of investigational therapeutic agents or enrollment in another therapeutic clinical trial at any institution. A minimum of 14 days or five half-lives of the drug (whichever is shorter) washout prior to start of daratumumab.
6. Refusal to participate in the long-term follow-up protocol.
7. Patients with active Central Nervous System (CNS) involvement by malignancy on magnetic resonance imaging (MRI) or by lumbar puncture.

   a. Patients with prior CNS disease that has been effectively treated will be eligible providing last treatment was ≥2 weeks before start of daratumumab and a remission documented within four weeks of planned CAR T-cell infusion by MRI brain and Cerebrospinal Fluid (CSF) analysis.
8. Previous recipients of allogeneic hematopoietic stem cell transplantation (AHCT) are excluded if they are <6 months post-transplant, have evidence of active graft-versus-host-disease (GVHD) of any grade, or are currently on immunosuppression.
9. Plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome, and AL amyloidosis.
10. Prior treatment with gene therapy or any gene-modified cellular therapy.
11. Cytotoxic chemotherapy, oral chemotherapeutic agents, or antibody-directed treatment within 14 days of starting daratumumab or after starting daratumumab.

    1. Corticosteroids are allowable up until seven days prior to starting daratumumab and after starting daratumumab for disease control up until the day prior to cell infusion (Day -1).
    2. Radiation is allowed to a single symptomatic site.
12. Patients post solid organ transplant who develop high-grade lymphomas or leukemias.
13. Concurrent active malignancy other than basal or squamous cell carcinomas of the skin.
14. Active bacterial, viral, or fungal infection requiring systemic treatment.
15. Patients who have received major surgery one week prior to starting daratumumab and three weeks prior to lymphodepletion.
16. Active malignancy that required therapy in the last two years except successfully treated non-metastatic basal or squamous cell carcinoma, or prostate carcinoma that does not require therapy. Other similar conditions may be discussed with and permitted by the medical monitor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade 3 or higher adverse events | start of therapy through 30 days after the end of study therapy, up to 2 years
  This measure is the number of Grade 3 or higher adverse events possibly, probably, or definitely related to the study therapy. Adverse events will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. Cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) will be graded and assessed using the American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading systems. Immune effector cell-associated hemophagocytic lymphohistiocytosis-like syndrome (IEC-HS) will be graded and assessed using the ASTCT panel guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Binod Dhakal, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No